CLINICAL TRIAL: NCT00914576
Title: Effect of Antioxidants on Oxygen Induced Vasoconstriction in LPS Induced Inflammatory Model in Humans
Brief Title: Effect of Antioxidants on Oxygen Induced Vasoconstriction in Lipopolysaccharide (LPS) Induced Inflammatory Model in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: OPHT-101108
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: Endotoxin, Escherichia Coli; Retina; Regional Blood Flow
MeSH Terms: conditions — Escherichia coli Infections | interventions — Vitamins; Oxygen; endotoxin, Escherichia coli; Lipopolysaccharides

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Vitamin and mineral supplement; Drug: 100% Oxygen; Drug: Escherichia coli Endotoxin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: 100% Oxygen; Drug: Escherichia coli Endotoxin

INTERVENTIONS:
Drug: Vitamin and mineral supplement — 1 capsule/day in the morning for 14 days, containing: Lutein 12mg, Vitamin C 300mg, Zinc 10mg, Ginko Biloba 10mg, Flavonoids 25mg, Fish oil 300mg
  Other Names: Vitamac Day
  Arms: 1
Drug: Vitamin and mineral supplement — 1 capsule/day in the evening for 14 days, containing: Zeaxanthin 5mg, Vitamin E 60mg, Copper 1mg, Selene 20µg, Ginko Biloba 10mg, Flavonoids 25mg, Alpha Lipon acid: 150mg
  Arms: 1
Drug: Placebo — 2 capsules/day for 14 days
  Arms: 2
Drug: 100% Oxygen — breathing of 100% O2 for 30 minutes on both study days
Drug: Escherichia coli Endotoxin — Escherichia coli Endotoxin (LPS, US Standard Reference Endotoxin, dose: 2 ng/kg bodyweight (corresponding to 20 IU/kg), i.v. bolus on both study days.
  Other Names: LPS (US Standard)

SUMMARY:
Oxidative stress has been implicated in playing a pathogenic role in many disease processes, especially in age-related disorders. It has been hypothesized that antioxidative agents such as vitamins and minerals, which are capable of scavenging free radicals, may reduce oxidative stress and may, in turn, be beneficial for patients with age-related disorders. Based on this hypothesis, several different combinations of vitamins have been introduced, all targeting at reducing oxidative stress. However, the in-vivo determination of the antioxidative properties of a certain drug or vitamin combination are hard to determine. In the current study, the researchers propose to investigate the effect of VITAMAC®, a combination of vitamins and minerals, in a systemic in-vivo inflammation model.

In the present study, the infusion of LPS, which is a cell wall component of Gram-negative bacteria and a major mediator in the pathogenesis of septic shock, will be used as a standardized experimental model of systemic inflammation in humans. Given that inflammation is associated with enhanced oxidative stress and widespread endothelial dysfunction, the LPS model is well suitable for determination of the antioxidative effects of VITAMAC®. As a main outcome parameter, the vascular reactivity of retinal vessels to systemic hyperoxia (induced by breathing 100% oxygen) will be tested in presence or absence of the antioxidant combination.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile (Must et al. 1991)
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 3 Dpt

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug, vitamins and minerals supplements as well
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Retinal blood flow | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhofer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Told R, Schmidl D, Palkovits S, Boltz A, Gouya G, Wolzt M, Witkowska KJ, Popa-Cherecheanu A, Werkmeister RM, Garhofer G, Schmetterer L. Antioxidative capacity of a dietary supplement on retinal hemodynamic function in a human lipopolysaccharide (LPS) model. Invest Ophthalmol Vis Sci. 2014 Dec 18;56(1):403-11. doi: 10.1167/iovs.14-15581. PMID 25525163
- [Derived] Told R, Palkovits S, Schmidl D, Boltz A, Gouya G, Wolzt M, Napora KJ, Werkmeister RM, Popa-Cherecheanu A, Garhofer G, Schmetterer L. Retinal hemodynamic effects of antioxidant supplementation in an endotoxin-induced model of oxidative stress in humans. Invest Ophthalmol Vis Sci. 2014 Apr 7;55(4):2220-7. doi: 10.1167/iovs.13-13784. PMID 24576874